CLINICAL TRIAL: NCT04189159
Title: PROMPT to Improve Speech Motor Abilities in Children With Cerebral Palsy
Brief Title: Speech Motor Treatment in Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Fondazione Stella Maris (Other)
Responsible Party: Principal Investigator, Simona Fiori, Principal Investigator, IRCCS Fondazione Stella Maris
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PROMPT-2019; 2019 Motor Speech Grant (Other Grant/Funding Number: The PROMPT Institute)
Record Dates: First submitted 2019-12-04; First posted 2019-12-06 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Cerebral Palsy; Dysarthria
Keywords: cerebral palsy; dysartria; motor speech treatment; prompt
MeSH Terms: conditions — Cerebral Palsy; Dysarthria

STUDY DESIGN:
Intervention Model Description: We plan a randomized trial using a wait-list control group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PROMPT Treated (Experimental): PROMPT treatment, twice a day, for 5 days a week, for 3 consecutive weeks
  Interventions: Behavioral: PROMPT
- Control (No Intervention): Usual treatment

INTERVENTIONS:
Behavioral: PROMPT — PROMPT treatment is consistent with the principles of motor learning, in that every session includes a blocked pre-practice followed by variable and distributed practice and a gradual, hierarchical increase of complexity. Speech motor goals are integrated in goals for language and functional communication. During a PROMPT session tactile-kinesthetic-proprioceptive inputs are consistently provided, in order to shape speech movements, to give information on sequencing and timing and to introduce constraints for the reduction of degrees of freedom at the articulators' level in favour of motor control.
  Other Names: motor speech treatment
  Arms: PROMPT Treated

SUMMARY:
Cerebral palsy (CP) is the most frequent cause of motor disability worldwide, with a prevalence of 2-2.5 per 1000 live births. Children with CP may experience a variety of difficulties with communication including speech. Communication impairment has been identified in at least 40% of children with CP, with 36-90% of CP children experiencing motor speech impairment.

The aims of the current project are to test the effectiveness of intensive PROMPT treatment in a group of preschool children with CP and motor speech disorders (dysarthria/apraxia of speech) and to evaluate differences to the intervention response according to CP type, brain lesion severity and white matter integrity of corticospinal tract. We hypothesize that children with CP and motor speech disorders will benefit from 3 weeks of daily administration of PROMPT treatment and show measurable improvement of speech intelligibility on clinical and kinematic assessments, with 3 months stability. Outcome measures will include a standardized speech motor assessment as well as improvement in kinematic speech measures detected by a computerized system. We also hypothesize that children with dyskynetic CP will show more improvement induced by the PROMPT treatment as compared to children with spastic CP. We finally hypothesize that corticospinal microstructural integrity positively impact on intelligibility recovery, with children with better integrity having bigger improvements.

Our study of PROMPT with children with varying types of CP meets current international priorities of testing and implementing effective, earlier interventions, therefore investing in the improvement infant's health based on evidence, as a future investment for individuals and the community.

DETAILED DESCRIPTION:
1. Rationale and purpose of research Cerebral palsy (CP) is the most frequent cause of motor disability worldwide, with a prevalence of 2-2.5 per 1000 live births. Several comorbidities characterize the clinical picture of children with CP, such as communication impairment, feeding difficulties, intellectual disability, vision and hearing impairment and epilepsy. Children with CP may experience a variety of difficulties with communication including speech, the development of gesture and facial expression, or receptive and expressive language, including voice production and intelligibility. Communication impairment has been identified in at least 40% of children with CP, with 36-90% of CP children experiencing motor speech impairment. Also, it has also been suggested that some children who do not present explicit dysarthria may have underlying speech motor control deficits. Intelligibility due to motor speech impairments affects activity and participation within various environments, reduces quality of life and increases daily care needs. Dysarthria may also be associated with excessive drooling and swallowing difficulties. Several studies consider compromised speech abilities as an indicator of the need for augmentative and alternative communication to supplement or replace communication. Conversely, CP and early acquired brain injury remain two of the most common medical causes of referral to speech and language therapy. However, little effort has been made in systematically improving speech motor abilities of children with CP by using early, reproducible and targeted intervention strategies. Furthermore, a poor relationship between the motor command and perceptual consequence of the speech movement has been hypothesized as a possible mechanism of speech dysfunction in CP, suggesting a potential therapeutic value of enhancing tactile-kinesthetic input to motor speech abilities of CP children.
2. Review of literature There are few papers reporting trials on targeted standardized intervention for speech motor deficit in infants or children with CP, with little evidences on treatment effectiveness. In a small group of children aged 3-11 years, it has been suggested that the effect of a speech motor treatment was aligned with the core principles of dynamic systems theory such as PROMPT (Prompts for Restructuring Oral Muscular Phonetic Targets) in changing speech motor patterns of children with CP with proven benefits in intelligibility, documented by kinematic analyses. Several types of CP were included (dyskinetic, spastic unilateral and bilateral). In a group of 7 children with spastic quadriplegia, some outcome of a motor speech treatment originally developed for adults with Parkinson disease were validated, the Lee Silverman Voice Treatment (LSVT LOUD). They also showed changes in white matter integrity supporting behavioral changes.
3. Research questions/Hypothesis Aim 1: To test the effectiveness of intensive PROMPT treatment in a group of preschool children with CP and motor speech disorders (dysarthria/apraxia of speech).

   Aim 2: To evaluate differences to the intervention response according to CP type, brain lesion severity and white matter integrity of corticospinal tract.

   Primary Hypothesis: children with CP and motor speech disorders will benefit from 3 weeks of daily administration of PROMPT treatment and show measurable improvement of speech intelligibility on clinical and kinematic assessments, with 3 months stability.

   Secondary hypotheses: children with dyskynetic CP will show more improvement induced by the PROMPT treatment as compared to children with spastic CP. Investigators also hypothesize that children with less severe brain lesions will have a higher level of improvement compared to children with more severe brain lesions. Investigators finally hypothesize that corticospinal microstructural integrity positively impact on intelligibility recovery, with children with better integrity having bigger improvements.
4. Method Investigators plan a randomized trial of PROMPT in children with CP using a wait-list control group. Eligible children will be randomized into either immediate treatment or wait-list-control groups. This design allows every child meeting inclusion criteria to eventually receive the treatment and avoids issues of equipoise. For CP wait-listed controls, the study continues for 3 weeks longer and results into an additional assessment.

Because PROMPT has been shown to be beneficial in several older children with CP, investigators' rational for the design allows for achievement of the RCT data collection and analysis, as well as allow all identified and consented children to receive the intervention.

The participants will include children between 3 and 9 years of age, with a diagnosis of CP and speech motor disorders. Parents will be asked to consent for the children for the participation in the study. All study activities will be carried out in our clinical center setting with a PROMPT trained therapist with appropriate knowledge of clinical research process.

In investigators' studies of rehabilitation with the CP population consent to participate in studies approaches 90%. From investigators' experience and clinical demographics of the center, they were expected 30 patients diagnosed CP with speech difficulties in the requisite age group per year, making possible a design of staggered enrollment of intervention and wait-list-control groups in the RCT. Recruitment will be completed according to the standards of research consent, followed by group randomization, by a team member other than the treating therapist. The assessments will be completed by an experiences SLP, different from the treating therapist.

ELIGIBILITY:
Inclusion Criteria:

* child between 2 and 9 years with a diagnosis of CP, with normal to mild intellectual disability and adequate language comprehension skills
* motor speech deficit

Exclusion Criteria:

* utilization of AAC strategies as the only means of communication,
* medical fragility or anatomical malformations affecting speech production preventing the ability to participate in the intervention

Ages: 2 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Verbal Motor Production Assessment for Children (VMPAC) | after the end of treatment period (4 weeks from baseline)
  Standardized motor speech assessment, which includes 5 subscales, where higher scores mean better performance: Global motor control (range 20-0); Focal oromotor control (range 268-0); Sequencing (range 46-0); Connected speech and language (range 45-0); Speech Characteristics (range 7-0)
Phonetic Inventory | after the end of treatment period (4 weeks from baseline)
  motor speech measure
the Intelligibility in Context Scale - Italian version | after the end of treatment period (4 weeks from baseline)
  motor speech measure, range 1-5, where higher scores mean better performances
Viking Speech Scale (VSS) | after the end of treatment period (4 weeks from baseline)
  Ordinal scale for intelligibility, range 1-4, with lower scores corresponding to better performances

SECONDARY OUTCOMES:
kinematic speech motor measures | after the end of treatment period (4 weeks from baseline)
  A kinematic analysis of facial movements during simple speech repetition tasks

CONTACTS AND LOCATIONS:
Overall Officials: Simona Fiori, MD, PhD, Principal Investigator — IRCCS Stella Maris Foundation
Locations (1):
- IRCCS Fondazione Stella Maris, Tirrenia, Tuscany, Italy

REFERENCES:
- [Background] Whelan MA. Practice parameter: diagnostic assessment of the child with cerebral palsy: report of the Quality Standards Subcommittee of the American Academy of Neurology and the Practice Committee of the Child Neurology Society. Neurology. 2004 Nov 23;63(10):1985-6; author reply 1985-6. No abstract available. PMID 15568275
- [Background] Barty E, Caynes K, Johnston LM. Development and reliability of the Functional Communication Classification System for children with cerebral palsy. Dev Med Child Neurol. 2016 Oct;58(10):1036-41. doi: 10.1111/dmcn.13124. Epub 2016 Apr 17. PMID 27087436
- [Background] Boliek CA, Fox CM. Therapeutic effects of intensive voice treatment (LSVT LOUD(R)) for children with spastic cerebral palsy and dysarthria: A phase I treatment validation study. Int J Speech Lang Pathol. 2017 Dec;19(6):601-615. doi: 10.1080/17549507.2016.1221451. Epub 2016 Oct 5. PMID 27705010
- [Background] Bosanquet M, Copeland L, Ware R, Boyd R. A systematic review of tests to predict cerebral palsy in young children. Dev Med Child Neurol. 2013 May;55(5):418-26. doi: 10.1111/dmcn.12140. PMID 23574478
- [Background] Chen CY, Liu CY, Su WC, Huang SL, Lin KM. Factors associated with the diagnosis of neurodevelopmental disorders: a population-based longitudinal study. Pediatrics. 2007 Feb;119(2):e435-43. doi: 10.1542/peds.2006-1477. PMID 17272605
- [Background] Cicchetti D. Neural plasticity, sensitive periods, and psychopathology. Dev Psychopathol. 2015 May;27(2):319-20. doi: 10.1017/S0954579415000012. No abstract available. PMID 25997757
- [Background] Cockerill H, Elbourne D, Allen E, Scrutton D, Will E, McNee A, Fairhurst C, Baird G. Speech, communication and use of augmentative communication in young people with cerebral palsy: the SH&PE population study. Child Care Health Dev. 2014 Mar;40(2):149-57. doi: 10.1111/cch.12066. Epub 2013 May 9. PMID 23656274
- [Background] Fiori S, Cioni G, Klingels K, Ortibus E, Van Gestel L, Rose S, Boyd RN, Feys H, Guzzetta A. Reliability of a novel, semi-quantitative scale for classification of structural brain magnetic resonance imaging in children with cerebral palsy. Dev Med Child Neurol. 2014 Sep;56(9):839-45. doi: 10.1111/dmcn.12457. Epub 2014 Apr 19. PMID 24750109
- [Background] Fiori S, Guzzetta A. Plasticity following early-life brain injury: Insights from quantitative MRI. Semin Perinatol. 2015 Mar;39(2):141-6. doi: 10.1053/j.semperi.2015.01.007. PMID 25813668
- [Background] Hustad KC, Gorton K, Lee J. Classification of speech and language profiles in 4-year-old children with cerebral palsy: a prospective preliminary study. J Speech Lang Hear Res. 2010 Dec;53(6):1496-513. doi: 10.1044/1092-4388(2010/09-0176). Epub 2010 Jul 19. PMID 20643795
- [Background] Kennes J, Rosenbaum P, Hanna SE, Walter S, Russell D, Raina P, Bartlett D, Galuppi B. Health status of school-aged children with cerebral palsy: information from a population-based sample. Dev Med Child Neurol. 2002 Apr;44(4):240-7. doi: 10.1017/s0012162201002018. PMID 11995892
- [Background] Liegeois F, Tournier JD, Pigdon L, Connelly A, Morgan AT. Corticobulbar tract changes as predictors of dysarthria in childhood brain injury. Neurology. 2013 Mar 5;80(10):926-32. doi: 10.1212/WNL.0b013e3182840c6d. Epub 2013 Feb 6. PMID 23390172
- [Background] McLeod S, Harrison LJ, McCormack J. The intelligibility in Context Scale: validity and reliability of a subjective rating measure. J Speech Lang Hear Res. 2012 Apr;55(2):648-56. doi: 10.1044/1092-4388(2011/10-0130). Epub 2012 Jan 3. PMID 22215036
- [Background] Mei C, Reilly S, Reddihough D, Mensah F, Pennington L, Morgan A. Language outcomes of children with cerebral palsy aged 5 years and 6 years: a population-based study. Dev Med Child Neurol. 2016 Jun;58(6):605-11. doi: 10.1111/dmcn.12957. Epub 2015 Nov 14. PMID 26566585
- [Background] Nordberg A, Miniscalco C, Lohmander A, Himmelmann K. Speech problems affect more than one in two children with cerebral palsy: Swedish population-based study. Acta Paediatr. 2013 Feb;102(2):161-6. doi: 10.1111/apa.12076. Epub 2012 Nov 27. PMID 23186066
- [Background] Novak I. Evidence-based diagnosis, health care, and rehabilitation for children with cerebral palsy. J Child Neurol. 2014 Aug;29(8):1141-56. doi: 10.1177/0883073814535503. Epub 2014 Jun 22. PMID 24958005
- [Background] Novak I, Morgan C, Adde L, Blackman J, Boyd RN, Brunstrom-Hernandez J, Cioni G, Damiano D, Darrah J, Eliasson AC, de Vries LS, Einspieler C, Fahey M, Fehlings D, Ferriero DM, Fetters L, Fiori S, Forssberg H, Gordon AM, Greaves S, Guzzetta A, Hadders-Algra M, Harbourne R, Kakooza-Mwesige A, Karlsson P, Krumlinde-Sundholm L, Latal B, Loughran-Fowlds A, Maitre N, McIntyre S, Noritz G, Pennington L, Romeo DM, Shepherd R, Spittle AJ, Thornton M, Valentine J, Walker K, White R, Badawi N. Early, Accurate Diagnosis and Early Intervention in Cerebral Palsy: Advances in Diagnosis and Treatment. JAMA Pediatr. 2017 Sep 1;171(9):897-907. doi: 10.1001/jamapediatrics.2017.1689. PMID 28715518
- [Background] Parkes J, Hill N, Platt MJ, Donnelly C. Oromotor dysfunction and communication impairments in children with cerebral palsy: a register study. Dev Med Child Neurol. 2010 Dec;52(12):1113-9. doi: 10.1111/j.1469-8749.2010.03765.x. Epub 2010 Aug 31. PMID 20813020
- [Background] Pennington L, Roelant E, Thompson V, Robson S, Steen N, Miller N. Intensive dysarthria therapy for younger children with cerebral palsy. Dev Med Child Neurol. 2013 May;55(5):464-71. doi: 10.1111/dmcn.12098. Epub 2013 Feb 26. PMID 23441834
- [Background] Pennington L, Parker NK, Kelly H, Miller N. Speech therapy for children with dysarthria acquired before three years of age. Cochrane Database Syst Rev. 2016 Jul 18;7(7):CD006937. doi: 10.1002/14651858.CD006937.pub3. PMID 27428115
- [Background] Ramig LO, Sapir S, Countryman S, Pawlas AA, O'Brien C, Hoehn M, Thompson LL. Intensive voice treatment (LSVT) for patients with Parkinson's disease: a 2 year follow up. J Neurol Neurosurg Psychiatry. 2001 Oct;71(4):493-8. doi: 10.1136/jnnp.71.4.493. PMID 11561033
- [Background] Reed A, Cummine J, Bakhtiari R, Fox CM, Boliek CA. Changes in White Matter Integrity following Intensive Voice Treatment (LSVT LOUD(R)) in Children with Cerebral Palsy and Motor Speech Disorders. Dev Neurosci. 2017;39(6):460-471. doi: 10.1159/000478724. Epub 2017 Jul 28. PMID 28750368
- [Background] Ward R, Strauss G, Leitao S. Kinematic changes in jaw and lip control of children with cerebral palsy following participation in a motor-speech (PROMPT) intervention. Int J Speech Lang Pathol. 2013 Apr;15(2):136-55. doi: 10.3109/17549507.2012.713393. Epub 2012 Oct 1. PMID 23025573
- [Background] Ward R, Leitao S, Strauss G. An evaluation of the effectiveness of PROMPT therapy in improving speech production accuracy in six children with cerebral palsy. Int J Speech Lang Pathol. 2014 Aug;16(4):355-71. doi: 10.3109/17549507.2013.876662. Epub 2014 Feb 13. PMID 24521506
- [Background] Watson RM, Pennington L. Assessment and management of the communication difficulties of children with cerebral palsy: a UK survey of SLT practice. Int J Lang Commun Disord. 2015 Mar-Apr;50(2):241-59. doi: 10.1111/1460-6984.12138. Epub 2015 Feb 4. PMID 25652139
- [Derived] Fiori S, Ragoni C, Podda I, Chilosi A, Amador C, Cipriani P, Guzzetta A, Sgandurra G. PROMPT to improve speech motor abilities in children with cerebral palsy: a wait-list control group trial protocol. BMC Neurol. 2022 Jul 6;22(1):246. doi: 10.1186/s12883-022-02771-6. PMID 35794522